CLINICAL TRIAL: NCT01538589
Title: Special Survey for Type 1 or Type 2 Diabetic Patients
Brief Title: Special Survey for Patients With Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1943
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin aspart users
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Prescribed by the physicians as a result of normal clinical practice

SUMMARY:
This study is conducted in Japan. The aim of this study is to evaluate the incidence of severe hypoglycaemia under normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no treatment history of insulin aspart (NovoRapid®)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes requiring insulin therapy with no treatment history of insulin aspart (NovoRapid®)
Sampling Method: Non-Probability Sample
Enrollment: 1582 (Actual)
Dates: Start 2003-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of severe hypoglycaemic symptoms | Year 1
Occurrence of severe hypoglycaemic symptoms | Year 2 for patients who had an antibody titre test performed
Antibody titre findings | Year 1
Antibody titre findings | Year 2 for patients who had an antibody titre test performed
Adverse events | Year 1
Adverse events | Year 2 for patients who had an antibody titre test performed

SECONDARY OUTCOMES:
Response rate assessed by the investigator: Ability or failure to achieve expected glycaemic control | Year 1
Response rate assessed by the investigator: Ability or failure to achieve expected glycaemic control | Year 2 for patients who had an antibody titre test performed
HbA1c (glycosylated haemoglobin) | Year 1
HbA1c (glycosylated haemoglobin) | Year 2 for patients who had an antibody titre test performed
Total dose of insulin infused subcutaneously | Year 1
Total dose of insulin infused subcutaneously | Year 2 for patients who had an antibody titre test performed

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com